CLINICAL TRIAL: NCT02562209
Title: To Determine the Effect of PACER Diet (High Protein Atkin's Complete VEgetaRian Diet) in Obese Subjects
Brief Title: High Protein Atkin's Complete (Lacto) VEgetaRian Diet (PACER) and Weight Loss
Acronym: PACER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diabetes Foundation, India (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Dr. Anoop Misra, Diabetes Foundation, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACER_2015
Record Dates: First submitted 2015-09-26; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Obesity
Keywords: Obesity; Abdominal adiposity; High protein diet
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PACER diet (Experimental): High Protein Atkin's Complete (Lacto) VEgetaRian Diet (PACER Diet) to be followed for 8 weeks.
  Interventions: Dietary Supplement: PACER Diet
- Standard weight reducing diet (Active Comparator): This group was prescribed Standard weight reducing diet to be followed for 8 weeks.
  Interventions: Other: Standard weight reducing diet

INTERVENTIONS:
Dietary Supplement: PACER Diet — Pacer diet to be followed for 8 weeks
  Arms: PACER diet
Other: Standard weight reducing diet — Standard weight reducing diet to be followed for 8 weeks
  Arms: Standard weight reducing diet

SUMMARY:
This study evaluates the effects "High Protein Atkin's Complete (lacto) VEgetaRian Diet (Acronym; 'PACER' diet) on weight, body composition and metabolic profiles in obese Asian Indians subjects living in north India.

DETAILED DESCRIPTION:
Increasing the protein consumption promotes weight loss through several mechanisms. Diets high in protein promote energy expenditure through increased postprandial thermogenesis, increase total daily expenditure and increase satiety as compared to carbohydrate. The present study aims to evaluate the effects "High Protein Atkin's Complete (lacto) VEgetaRian Diet (Acronym; 'PACER' diet) on weight, body composition and metabolic profiles in obese Asian Indians subjects living in north India.

ELIGIBILITY:
Inclusion Criteria

* Age 25 to 60 years
* Body mass index (BMI) ≥ 25 kg/m2 to 40 kg/m2
* Subjects who have stable weight, i.e. who have not had more than ± 3 kg variation in their weight level in the 3 months prior to screening for this study.
* Absence of significant disease or clinically significant medical history or physical examination during screening in the view of the investigator.
* Subjects willing to provide written inform consent to participate in the study.

Exclusion Criteria

* Body mass index (BMI) > 40 kg/m2
* Any patient taking/requiring drugs known to effect insulin resistance, lipids, vascular reactivity, during the intervention period would be excluded from the study
* Patients on any drugs that change the weight or in conditions where dietary protein supplementation is contraindicated
* Subjects who are consuming a high protein diet on randomization, to be excluded
* Acute infections or chronic debilitating diseases like tuberculosis, malignancy, HIV infection etc
* Any life threatening serious disorder of the liver, kidneys, heart, lungs or other organs
* Pregnancy & lactation
* Patients having diagnosed with any of the following:

  * Type 2 diabetes mellitus
  * Cushing's disease
  * Severe end organ damage
* Unwillingness to give written informed consent for participation in the study

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2012-01; Primary Completion 2014-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Weight loss (kg) | 8 weeks

SECONDARY OUTCOMES:
Lipid profile | 8 weeks
Insulin resistance | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — Diabetes Foundation, India
Locations (1):
- Fortis Flt Lt Rajan Dhall Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Background] Bhardwaj S, Misra A. Obesity, diabetes and the Asian phenotype. World Rev Nutr Diet. 2015;111:116-22. doi: 10.1159/000362308. Epub 2014 Nov 17. No abstract available. PMID 25418400
- [Background] Jenkins DJ, Wong JM, Kendall CW, Esfahani A, Ng VW, Leong TC, Faulkner DA, Vidgen E, Greaves KA, Paul G, Singer W. The effect of a plant-based low-carbohydrate ("Eco-Atkins") diet on body weight and blood lipid concentrations in hyperlipidemic subjects. Arch Intern Med. 2009 Jun 8;169(11):1046-54. doi: 10.1001/archinternmed.2009.115. PMID 19506174